CLINICAL TRIAL: NCT04975776
Title: Sleep Restriction Therapy for Insomnia Delivered as Group Therapy in Primary Health Care: A Randomized Controlled Trial
Brief Title: Sleep Restriction Therapy for Insomnia in Primary Health Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FoUI-936149
Record Dates: First submitted 2021-07-15; First posted 2021-07-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Insomnia
Keywords: Disorders of Initiating and Maintaining Sleep; DIMS; Early Awakening; Awakening, Early; Nonorganic Insomnia; Insomnia, Nonorganic; Primary Insomnia; Insomnia, Primary; Transient Insomnia; Insomnia, Transient; Rebound Insomnia; Insomnia, Rebound; Secondary Insomnia; Insomnia, Secondary; Sleep Initiation Dysfunction; Dysfunction, Sleep Initiation; Dysfunctions, Sleep Initiation; Sleep Initiation Dysfunctions; Sleeplessness; Insomnia Disorder; Insomnia; Insomnias; Chronic Insomnia; Insomnia, Chronic; Psychophysiological Insomnia; Insomnia, Psychophysiological
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A multi-center randomized controlled trial in primary health care with two parallel study arms: (1) sleep restriction group therapy (experimental condition) and (2) sleep hygiene (control condition).
Who Masked: Investigator
Masking Description: Study staff entering data will be blinded to the condition. The researchers will provide some supervision to the health care professional who deliver the treatment. The researchers will therefore know the identities of the health care professionals they supervise. However, outcome data will be pseudonymized, so researchers will be blinded during outcome assessment. It is not possible to blind the health care professionals delivering the treatment or patients receiving it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep restriction therapy (Experimental): Four group sessions delivered at the participants' primary health care centers once a week for 3 weeks and again after a 4-week pause. The first session will last for 2 hours and the other sessions for 1 hour.
  Interventions: Behavioral: Sleep restriction therapy
- Sleep hygiene (Active Comparator): Participants in the active comparator group will receive a brochure with sleep hygiene advice from the primary health care center at baseline.
  Interventions: Behavioral: Sleep hygiene

INTERVENTIONS:
Behavioral: Sleep restriction therapy — The intervention includes psychoeducation and sleep restriction therapy, sleep restriction instructions, problem-solving, and support for participants in adjusting sleep restriction instructions to their individual needs and life circumstances. At the final session, participants create an individual plan for maintaining new sleep habits and coping with insomnia relapse. During the intervention, participants are free to seek and receive standard care for insomnia.
  Arms: Sleep restriction therapy
Behavioral: Sleep hygiene — The control condition will include written, general information about sleep and lifestyle and environmental factors that could improve or disturb sleep. The participants will be free to seek and receive standard care for insomnia.
  Arms: Sleep hygiene

SUMMARY:
The recommended treatment for insomnia, cognitive behavioral therapy for insomnia (CBT-I), is effective. However, its long, multi-component nature makes it challenging to implement in ordinary primary care, where most people are treated. An important component of CBT-I is sleep restriction therapy, which may be comparatively easy to carry out in routine primary care. This project tests whether a brief nurse-led group intervention in primary care based on sleep restriction therapy for insomnia reduces insomnia severity and is cost-effective.

DETAILED DESCRIPTION:
Background: Insomnia is typically treated in primary health care. The most common treatment is hypnotic drugs, despite their limited and short-term effects, the risk for adverse side effects and dependence, and the fact that CBT-I is the recommended first-line treatment. Reasons may include lack of knowledge about insomnia, a culture of prescribing hypnotics, lack of time during consultations, and a shortage of CBT-I providers. Sleep restriction therapy is one of the core components of CBT-I. It is a behavioral technique that may be feasible to deliver in routine care with existing resources and time constraints.

Objectives: This randomized controlled trial aims to investigate whether brief, behavioral group therapy in primary care based on sleep restriction therapy reduces insomnia severity and is cost-effective. A process evaluation will explore barriers and facilitators for participation and delivery.

Methods: Health care professionals from participating primary health care centers will complete a 1.5-day digital course on assessing patients for insomnia and delivering the intervention. Patients who seek primary health care and meet the study criteria will be randomized to sleep restriction therapy or to receive written sleep hygiene information. Both groups will be free to seek and receive standard care for insomnia. Sociodemographic and clinical characteristics will be collected prior to baseline. Study outcomes include insomnia severity, sleep, daytime symptoms, quality of life, use of hypnotics, sick leave, and work ability. Outcomes will be assessed over a 24-month period. The cost-effectiveness analysis will include the number of insomnia-free days at the 12-month follow-up and quality-adjusted life years. Patient characteristics will be analyzed in relation to adherence, and response. Qualitative explorations of patients and nurses' experiences will be conducted alongside the trial (approximately 15 patients and 15 nurses).

ELIGIBILITY:
Inclusion Criteria:

* Fulfills the DSM-5 diagnostic criteria for insomnia disorder: a) Difficulty initiating sleep, difficulty maintaining sleep, and early morning awakenings despite adequate opportunity for sleep (e.g., adequate time and circumstances for sleep and a safe, quiet, and dark bedroom). b) The sleep difficulties cause significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning. c) The sleep difficulties occur at least 3 nights per week and have been present for at least 3 months. d) The symptoms are not better explained by and do not occur exclusively during the course of another sleep-wake disorder. e) The symptoms cannot be attributed to the effects of a substance (e.g., drug abuse and medication). f) Coexisting mental disorders and medical conditions do not adequately explain the predominant complaint of insomnia.

Exclusion Criteria:

* Severe psychiatric illness (e.g., severe depression, schizophrenia, bipolar disorder)
* Suicidal ideation
* Untreated sleep disorder other than insomnia (e.g., sleep apnea, and restless legs syndrome)
* Epilepsy
* Cognitive disorder
* Pregnancy
* Night shift work
* Language difficulties (inability to understand and speak Swedish well enough to participate in the intervention and respond to measurement instruments)
* ≤ 7 points on the Insomnia Severity Index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) score | Baseline and 3, 6, 12, and 24 months after baseline
  The ISI is a 7-item scale that asesses the severity of sleep disturbance, how much sleep disturbance interferes with daily life and functioning, the noticeability of these impairments to others, worry and distress resulting from sleep disturbance, and general sleep satisfaction/dissatisfaction. Responses are provided on a Likert-scale (0-4). The total score ranges from 0 to 28, and higher scores indicate more severe problems.

SECONDARY OUTCOMES:
Change in sleep efficiency derived from sleep diary | Baseline and 3, 12, and 24 months after baseline
  Sleep efficiency (percentage of time asleep while in bed) will be calculated on the basis of self-reported sleep at each measurement point.
Change in sleep onset latency derived from sleep diary | Baseline and 3, 12, and 24 months after baseline
  Sleep onset latency (time to initiation of sleep after going to bed for the night) will be calculated on the basis of self-reported sleep at each measurement point.
Change in time awake after sleep onset derived from sleep diary | Baseline and 3, 12, and 24 months after baseline
  Time awake after sleep onset calculated on the basis of self-reported sleep at each measurement point.
Change in number of nocturnal awakenings derived from sleep diary | Baseline and 3, 12, and 24 months after baseline
  Number of nocturnal awakenings calculated on the basis of self-reported sleep at each measurement point.
Change in sleep quality derived from sleep diary | Baseline and 3, 12, and 24 months after baseline
  Perceived sleep quality will be calculated on the basis of self-reported sleep at each measurement point. The variable is rated on a Likert scale ranging from 1 to 5. Higher scores indicate better sleep quality.
Change in Fatigue Severity Scale (FSS) score | Baseline and 3, 12, and 24 months after baseline
  The FSS is a 9-item scale that measures the interference of fatigue with daily life. Each item is rated on a scale that ranges from 1 to 7. Higher total scores indicate more severe fatigue.
Change in the Montgomery-Asberg Depression Rating Scale - self-rating version (MADRS-S) score | Baseline and 3, 12, and 24 months after baseline
  MADRS-S includes 9 items that measure the severity of depressive symptoms (mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism, and zest for life). Each item includes six statements ranging from the most positive (statement 0) to the least positive (statement 6). The total score ranges from 0 to 54. The higher the score, the more severe the symptoms.
Changes in the EQ-5D score | Baseline and 3, 12, and 24 months after baseline
  EQ-5D is a generic measure of health status that measures quality of life in five health domains: mobility, self-care, daily activities, pain/suffering, and anxiety/depression. The response scale for each domain ranges from no problems (0) to severe problems (3). EQ-5D also includes a visual scale for each theme and for overall health status. Together, the responses form 248 different health profiles, each of which is assigned a point value that makes it possible to compare results.
Changes in the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) score | Baseline and 3, 12, and 24 months after baseline
  DBAS measures dysfunctional beliefs and attitudes on an analog scale labeled "strongly disagree" to the left and "strongly agree" to the right. Respondents place a vertical mark at the point on the line that corresponds to degree that they disagree or agree with the statement. The distance (mm) from the left end of the line to the vertical mark is measured and used as the score. Scores range from 0 to 100. Higher scores indicate stronger agreement with the statement.
Changes in Work Ability Index (WAI) score | Baseline, 1 year after baseline, and 2 years after baseline
  The WAI includes seven domains that measure current work ability compared with the lifetime best (0-10 points), work ability in relation to the demands of the job (2-10 points), number of current diseases diagnosed by a physician (1-7 points), estimated work impairment due to diseases (1-6 points), sickness leave during the past year (1-5 points), own prognosis of work ability two years from now (1, 4, or 7 points), and mental resources (1-4 points). The total score ranges from 7 to 49. Higher scores indicate better work ability.
Changes in Short Form Health Survey-12 (SF- 12) score | Baseline and 3, 12, and 24 months after baseline
  The SF-12 includes 12 items that measure health-related quality of life. The number of response alternatives varies by item. An algorithm is used to calculate final scores, which range from 0 to 100. Higher score indicate better quality of life.
Change in Work and Social Adjustment Scale (WSAS) scores | Baseline and 3, 12, and 24 months after baseline
  The WSAI is a 5-item scale that measures functional impairment related to sleep problems. Response alternatives range from 0 (not at all) to 8 (very severely). The total score ranges from 0 to 40. Higher scores indicate more severe impairment.
Changes in self-reported hypnotic drug use | Baseline and 3, 12, and 24 months after baseline
  A questionnaire that measures the frequency (including name and amount taken) of the use of prescribed hypnotics on a Likert scale ranging from never (1) to daily (6). Higher scores indicate more frequent use.
Changes in self-reported sick leave | Baseline, 1 year after baseline, and 2 years after baseline
  Participants will be asked to report the number of days they have been on sick leave.
Treatment side effects | 3 months after baseline
  Participants will complete a questionnaire that includes 10 items that measure the perceived severity of potential side effects of sleep restriction therapy on a Likert scale. The scores range from 1 to 4. Higher scores indicate more severe side effects. The questionnaire also includes a question asking about the time for side effects (e.g., in the beginning of treatment, mid-treatment etc.).
Treatment adherence | 3 months after baseline
  Participants will complete a questionnaire that includes nine items that measure self-rated adherence to sleep restriction therapy on a Likert scale. Higher scores indicate better adherence. The score on each item range from 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Sandlund, PhD, Principal Investigator — Region Stockholm
Locations (1):
- Christina Sandlund, Stockholm, Stockholms Läns Landsting, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maurer LF, Schneider J, Miller CB, Espie CA, Kyle SD. The clinical effects of sleep restriction therapy for insomnia: A meta-analysis of randomised controlled trials. Sleep Med Rev. 2021 Aug;58:101493. doi: 10.1016/j.smrv.2021.101493. Epub 2021 Apr 21. PMID 33984745
- [Background] Kyle SD, Morgan K, Spiegelhalder K, Espie CA. No pain, no gain: an exploratory within-subjects mixed-methods evaluation of the patient experience of sleep restriction therapy (SRT) for insomnia. Sleep Med. 2011 Sep;12(8):735-47. doi: 10.1016/j.sleep.2011.03.016. Epub 2011 Sep 9. PMID 21907616
- [Background] Sandlund C, Hetta J, Nilsson GH, Ekstedt M, Westman J. Improving insomnia in primary care patients: A randomized controlled trial of nurse-led group treatment. Int J Nurs Stud. 2017 Jul;72:30-41. doi: 10.1016/j.ijnurstu.2017.03.007. Epub 2017 Apr 14. PMID 28445790
- [Background] Sandlund C, Kane K, Ekstedt M, Westman J. Patients' experiences of motivation, change, and challenges in group treatment for insomnia in primary care: a focus group study. BMC Fam Pract. 2018 Jul 9;19(1):111. doi: 10.1186/s12875-018-0798-2. PMID 29986651
- [Background] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- See also: Academic Primary Health Care Centre, Region Stockholm — https://www.akademisktprimarvardscentrum.se/om-oss/projektkatalog/forskning-for-att-effektivare-bedoma-och-behandla-somnproblem-i-primarvarden/